CLINICAL TRIAL: NCT00525733
Title: A Phase II, Randomized Trial of Open-Label Truvada With Darunavir/Ritonavir Versus Multiclass Therapy With Truvada, Darunavir/Ritonavir, Maraviroc and Raltegravir in Acutely HIV-1 Infected Antiretroviral-Naïve Subjects
Brief Title: Standard Antiretroviral v. Multi-class Therapy in Acutely HIV-1 Infected Antiretroviral-Naïve Subjects (ADARC 2007-01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Aaron Diamond AIDS Research Center (Other); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMA-0610-0607
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
Keywords: HIV-1; Acute Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Racivir; Maraviroc; Raltegravir Potassium; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-drug standard therapy (Active Comparator): FTC 200 mg/TDF 300 mg QD + darunavir 800 mg/ +ritonavir 100 mg QD
  Interventions: Drug: darunavir 800 mg; Drug: FTC 200 mg/TDF 300mg; Drug: Ritonavir 100 mg
- 5-drug experimental therapy (Experimental): FTC 200 mg/TDF 300 mg QD + darunavir 800 mg + ritonavir 100 mg QD + Raltegravir 400 mg BID + Maraviroc 150 mg BID
  Interventions: Drug: darunavir 800 mg; Drug: FTC 200 mg/TDF 300mg; Drug: Maraviroc; Drug: Raltegravir; Drug: Ritonavir 100 mg

INTERVENTIONS:
Drug: darunavir 800 mg — darunavir 800mg tablet will be administered with 100 mg capsule of ritonavir once daily (may be taken with or without food)
  Other Names: prezista
Drug: FTC 200 mg/TDF 300mg — Emtricitabine/tenofovir DF fixed-dose tablet containing 200 mg of emtricitabine and 300 mg of tenofovir DF will be administered orally as one tablet once daily (may be taken with or without food)
  Other Names: FTC/TDF
Drug: Maraviroc — Maraviroc will be administered twice daily in 150 mg tablets (may be taken with or without food)
  Other Names: selzentry
  Arms: 5-drug experimental therapy
Drug: Raltegravir — Raltegravir will be administered twice daily as 1-400 mg tablets (to be taken with food)
  Other Names: isentress
  Arms: 5-drug experimental therapy
Drug: Ritonavir 100 mg — one tablet of ritonavir is taken with darunavir daily
  Other Names: norvir

SUMMARY:
The researchers are involved in a phase II, randomized, two-arm study, comparing the efficacy, safety, and tolerability of open-label ritonavir (RTV)-enhanced darunavir with Truvada to a 5-drug multi-class regimen including truvada, darunavir/ritonavir/maraviroc/and raltegravir on acutely HIV-1-infected, antiretroviral (ARV) drug-naïve men and women. Subjects will participate for at least 60 weeks and up to 96 weeks if in the opinion of the investigator and patient that continued therapy is in the patient's best interest.

Hypotheses:

* Multi-class antiretroviral therapy (ART) is superior to RTV-enhanced ATV in combination with Emtricitabine/Tenofovir DF (FTC/TDF) with respect to suppression of viral replication.
* Multi-class ART is superior to RTV-enhanced ATV in combination with FTC/TDF with respect to immune reconstitution in peripheral blood and in the gastrointestinal mucosa.
* Multi-class ART is equivalent to RTV-enhanced ATV in combination with FTC/TDF with respect to tolerability.

DETAILED DESCRIPTION:
* DURATION: Subjects will participate for at least 60 weeks and up to 96 weeks if in the opinion of the investigator and patient that continued therapy is in the patient's best interest.
* SAMPLE SIZE: 36 subjects randomized 2:1 multi-class versus standard antiretroviral therapy.
* POPULATION: Acutely HIV-1-infected, antiretroviral (ARV) drug-naïve (≤ 7 days of ARV treatment at anytime prior to study entry*) men and women ≥ 18 years of age.
* REGIMEN: At entry subjects will be randomized to one of the following in a 1:2 ratio:

ARM A: FTC 200 mg/TDF 300 mg QD + darunavir 800 mg/ritonavir 100 mg QD

ARM B: FTC 200 mg/TDF 300 mg QD + darunavir 800mg/ritonavir 100 mg QD + Raltegravir 400 mg BID + Maraviroc 150 mg BID

The three primary objectives are:

1. To assess whether a multi-class regimen could completely suppress virus replication in HIV infected individuals based on:

   * Plasma HIV-1 RNA levels at 48 weeks
   * Ultrasensitive < 50 copy assay
   * 5 copy assay
   * 1 copy assay
   * Cell associated HIV-1RNA levels at week 48
   * Proviral DNA
   * Levels at week 48
   * Decay rates from week 12 to week 48
2. To determine whether multi-class antiviral therapy results in enhanced immune reconstitution in peripheral blood and gastrointestinal mucosa based on flow and immunohistochemistry.
3. To assess tolerability of multi-class compact antiviral therapy to that of standard compact antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute HIV-1 infection defined as:

  * Negative ELISA/Western Blot or indeterminate Western Blot in the presence of HIV-1 RNA > 5,000 copies/ml.
  * Positive HIV-1 serology with a detuned ELISA O.D. value below 0.5.
  * A documented negative serology within 180 days of screening and a positive HIV-1 serology at screening
* Antiretroviral (ARV) drug-naïve (defined as ≤ 7 days of ARV treatment at any time prior to entry*).
* The only exceptions are:

  * Use of antivirals as part of post-exposure prophylaxis (PEP) provided the subject did not acquire HIV-1 infection from the event that required PEP.
  * Therapy with an investigational ARV drug that was not an NRTI, NNRTI, or PI.
* Laboratory values obtained within 30 days prior to study entry.

  * Absolute neutrophil count (ANC) ≥ 500/mm3
  * Hemoglobin ≥ 8.0 g/dL
  * Platelet count ≥ 40,000/mm3
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 7.5 × ULN
  * Total bilirubin ≤2.5 x ULN
  * Calculated creatinine clearance ≥60 mL/min as estimated by the Cockcroft-

Gault equation:

For men, (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72) = CrCl (mL/min)*

* For women, multiply the result by 0.85 = CrCl (mL/min) NOTE: A program to assist in calculations is available on the DMC web site at: http://www.fstrf.org/ACTG/ccc.html
* For women of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to initiating study medications unless otherwise specified by product labeling.
* Female candidates of reproductive potential is defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) or have not undergone surgical sterilization (e.g., hysterectomy, or bilateral oophorectomy, or bilateral tubal ligation).

Contraception requirements:

* Female candidates of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree that they will use at least one reliable method of contraception while receiving the protocol-specified drugs and for 6 weeks after stopping the medications.

Male Candidates:

* If you are a heterosexual male, you and your sexual partner must agree to use acceptable methods of birth control during the entire study.
* Acceptable methods of birth control include intrauterine device (IUD), diaphragm with spermicide, condoms or not having sex.
* Oral contraceptives alone are not an acceptablemethod of birth control.
* Men and women age ≥ 18 years.
* Ability and willingness of subject to give written informed consent.

Exclusion Criteria:

* Currently breast-feeding.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. NOTE: Subjects receiving stable physiologic glucocorticoid doses, defined as prednisone ≤ 10 mg/day, will not be excluded.
* Known allergy/sensitivity to study drugs or their formulations.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry.

NOTE: Oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses (as judged by the site investigator) have no restriction.

* Clinically relevant cardiac conduction system disease. This includes severe first degree atrioventricular block (PR interval > 0.26 seconds), or second, or third-degree atrioventricular block.
* Requirement for any current medications that are prohibited with any study treatment.
* Evidence of major resistance-associated mutations on genotype performed within 14 days of day 1. Major resistance-associated mutations include: NRTI: K65R or inserts Q151M, M184V/I, PI: I50L/V, I84V, N88S.
* Viral population that is either dual tropic or X4 tropic using the Monogram assay (patients will be entered and be treated pending this result performed within 28 days of day 1).
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical (e.g., infectious disease) illness.
* Participation in any other clinical trial within 30 days prior to screening.
* Any other clinical conditions or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Principal Investigator — Rockefeller University
Locations (2):
- United States (2):
  - Rockefeller University, New York, New York
  - The Rockefeller University, New York, New York

REFERENCES:
- See also: The Rockefeller University Hospital — http://www.rucares.org/clinicalstudies/list.php?searchTerm=&x=20&y=12&pi_id=29

RESULTS

PARTICIPANT FLOW:
Groups:
- 3-drug Standard Therapy: FTC 200 mg/TDF 300 mg QD + darunavir 800 mg/ritonavir 100 mg QD
  darunavir: Darunavir 800mg tablet will be administered with 100 mg capsule of ritonavir once daily (may be taken with or without food)
  Emtricitabine/tenofovir DF: Emtricitabine/tenofovir DF fixed-dose tablet containing 200 mg of emtricitabine and 300 mg of tenofovir DF will be administered orally as one tablet once daily (may be taken with or without food)
- 5-drug Experimental Therapy: FTC 200 mg/TDF 300 mg QD + darunavir 800 mg/ritonavir 100 mg QD + Raltegravir 400 mg BID + Maraviroc 150 mg BID
  darunavir: Darunavir 800mg tablet will be administered with 100 mg capsule of ritonavir once daily (may be taken with or without food)
  Emtricitabine/tenofovir DF: Emtricitabine/tenofovir DF fixed-dose tablet containing 200 mg of emtricitabine and 300 mg of tenofovir DF will be administered orally as one tablet once daily (may be taken with or without food)
  Maraviroc: Maraviroc will be administered twice daily in 150 mg tablets (may be taken with or without food)
  Raltegravir: Raltegravir will be administered twice daily as 1-400 mg tablets (to be taken with food)
Period: Overall Study
Arm/Group | 3-drug Standard Therapy | 5-drug Experimental Therapy
Started | 14 | 26
Completed | 11 | 23
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: This is an as treated analysis. Baseline characteristics describe subjects available for primary endpoint analysis at week 48. There were 34 subjects available for primary endpoint analysis however 2 subjects were not able to be analyzed due to primer mismatch therefore results are available for 32 subjects in the primary endpoint analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3-drug Standard Therapy | 5-drug Experimental Therapy | Total
Number analyzed (Participants) | 11 | 23 | 34
Age, Continuous [Mean (Full Range); unit: years] | 37 [25 to 48] | 41 [29 to 69] | 38 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 23 | 34
Region of Enrollment [Number; unit: participants]
  United States | 11 | 23 | 34
Mean log baseline HIV-1 RNA [Mean (Full Range); unit: log copies/mL] | 5.6 [3.1 to 6.4] | 6.3 [4.8 to 7.0] | 5.8 [3.1 to 7.0]
Mean CD4+ T-cell count [Mean (Full Range); unit: cells/mm^3] | 539 [230 to 1066] | 405 [305 to 524] | 496 [230 to 1066]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome of This Study is the Proportion of Patients Having Detectable HIV-1 RNA Using the Single Copy Assay After 48 Weeks of Treatment and the Study Hypothesis is That New Treatment is Better Than the Control Group.
Time Frame: 48 weeks
Measure: Number; unit: # subjects without detectable viremia
Arm/Group | 3-drug Standard Therapy | 5-drug Experimental Therapy
Number analyzed (Participants) | 11 | 21
# subjects without detectable viremia | 3 | 9
Statistical Analysis 1: Comparison: 3-drug Standard Therapy vs 5-drug Experimental Therapy; Test type: Superiority or Other; p = 0.46, Chi-squared

ADVERSE EVENTS:
Arm/Group | 3-drug Standard Therapy | 5-drug Experimental Therapy
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/23
Other Adverse Events (participants affected / at risk) | 0/11 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes